CLINICAL TRIAL: NCT02649309
Title: Effect of Single-cycle Remote Ischemic Preconditioning and Postconditioning on Myocardial Injury in Patients Undergoing Emergency and Elective Percutaneous Intervention in Phramongkutklao Hospital and Thammasat University
Brief Title: Single-cycle Remote Ischemic Preconditioning and Postconditioning (SCRIP) Trial
Acronym: SCRIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: PMK-SCRIP
Record Dates: First submitted 2015-12-01; First posted 2016-01-07 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Reperfusion Injury
Keywords: Ischemic Preconditioning; Postconditioning; Angioplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RIPre + RIPost (Experimental): Intervention: RIPre 200 mmHg + RIPost 200 mmHg
  Interventions: Procedure: RIPre; Procedure: RIPost
- RIPre + Sham (Experimental): Intervention: RIPre 200 mmHg + Sham 10 mmHg
  Interventions: Procedure: RIPre; Procedure: Sham-Post
- Sham + RIPost (Experimental): Intervention: Sham 10 mmHg + RIPost 200 mmHg
  Interventions: Procedure: Sham-Pre; Procedure: RIPost
- Sham + Sham (Sham Comparator): Intervention: Sham 10 mmHg + Sham 10 mmHg
  Interventions: Procedure: Sham-Pre; Procedure: Sham-Post

INTERVENTIONS:
Procedure: RIPre — Preconditioning 200 mmHg x 5 minutes before procedure
  Arms: RIPre + RIPost; RIPre + Sham
Procedure: Sham-Pre — Sham 10 mmHg x 5 minutes before procedure
  Arms: Sham + RIPost; Sham + Sham
Procedure: RIPost — Postconditioning 200 mmHg x 5 minutes after procedure
  Arms: RIPre + RIPost; Sham + RIPost
Procedure: Sham-Post — Sham 10 mmHg x 5 minutes after procedure
  Arms: RIPre + Sham; Sham + Sham

SUMMARY:
This trial is a 2 x 2 factorial design, double-blinded, randomized controlled trial to evaluate efficacy and safety of remote ischemic preconditioning and postconditioning in patient undergoing coronary angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for percutaneous coronary intervention (elective and emergency cases)
* Age > 18-year-old
* Informed consent

Exclusion Criteria:

* Previous CABG
* Previous PCI in 1 week / treatment with thrombolysis within 30 days
* Peripheral arterial disease / A-V shunt of upper extremities (AVF for hemodialysis)
* Paresis of upper limb
* Unstable patient such as cardiogenic shock / vasopressor / IABP / cooling (hypothermia)
* Fatal cardiac arrhythmia (VT / VF)
* Chronic hypoxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac Troponin-T from baseline | within 24 hours

SECONDARY OUTCOMES:
Incidence of myocardial injury | within 24 hours
  Incidence of myocardial injury defined as > 5 times elevation of cardiac troponin from baseline in patients with normal baseline troponin and elevation of cardiac troponin > 20% in patients who have elevated baseline troponin (>99 percentile upper reference limit).
Major adverse cardiovascular events (MACE) in each intervention group | 6 months
  MACE = composite of CV death, MI, stroke, repeat revascularization, hospitalization for heart failure.
Incidence of myocardial injury in differrent subgroups of patient characteristics | within 24 hours
  Patient characteristics include sex, age, underlying disease, medications, indication for PCI (ACS and elective PCI), baseline cardiac enzyme and creatinine. Incidence of myocardial injury defined as > 5 times elevation of cardiac troponin from baseline in patients with normal baseline troponin and elevation of cardiac troponin > 20% in patients who have elevated baseline troponin (>99 percentile upper reference limit).
Incidence of myocardial injury in patients with vs. without RIPre and RIPost | 24 hours
  Myocardial injury defined as > 5 times elevation of cardiac troponin from baseline in patients with normal baseline troponin and elevation of cardiac troponin > 20% in patients who have elevated baseline troponin (>99 percentile upper reference limit).
Incidence of MACE in differrent subgroups of patient characteristics | 6 months
  Patient characteristics include sex, age, underlying disease, medications, indication for PCI (ACS and elective PCI), baseline cardiac enzyme and creatinine.
  MACE = composite of CV death, MI, stroke, repeat revascularization, hospitalization for heart failure.
Incidence of MACE in patients with vs. without RIPre and RIPost | 6 months
  Patient characteristics include sex, age, underlying disease, medications, indication for PCI (ACS and elective PCI), baseline cardiac enzyme and creatinine.
  MACE = composite of CV death, MI, stroke, repeat revascularization, hospitalization for heart failure.
Incidence of MACE in patients who have myocardial injury vs. patients who have no myocardial injury | 6 months
  Myocardial injury defined as > 5 times elevation of cardiac troponin from baseline in patients with normal baseline troponin and elevation of cardiac troponin > 20% in patients who have elevated baseline troponin (>99 percentile upper reference limit).

CONTACTS AND LOCATIONS:
Overall Officials: Nakarin Sansanayudh, MD,PhD, Principal Investigator — Department of Internal Medicine, Phramongkutklao Hospital, Bangkok, Thailand
Locations (1):
- Department of Internal Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes